CLINICAL TRIAL: NCT06230445
Title: A Phase 3, Randomized, Open-label Trial of Digital Therapeutic vs Regular Follow-up in Whole Process Management of Lung Cancer
Brief Title: Effects of Digital Therapeutic in Whole Process Management of Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hao Long, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A2023-002
Record Dates: First submitted 2023-08-31; First posted 2024-01-30 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Application of Digital Therapeutic in Lung Cancer Whole Process Management
Keywords: Digital therapeutic; Whole process management; Lung cancer; Patient follow-up
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UHealth digital therapeutic group (Experimental): The patients in this group will use UHealth application to monitor their symptoms and give medical advisement through digital methods.
  Interventions: Other: UHealth digital therapeutic
- Regular follow-up group (No Intervention): The patients in this group will use paper-based follow-up to monitor their symptoms and give medical advisement in outpatient clinic.

INTERVENTIONS:
Other: UHealth digital therapeutic — UHealth digital therapeutic is an application that patients can report their symptoms. If the contents that patients fill in reach the threshold, UHealth application will automatic report to doctor and the doctor will give medical advisement through UHealth digital therapeutic application.
  Arms: UHealth digital therapeutic group

SUMMARY:
This trial will randomize patients into two groups, the treatment group will use the digital therapeutic application named 'UHealth' for the whole process management and the control group will use regular follow-up. The trial aims to look into the difference between quality of life, anxiety/depression index, emergency treatment times, hospital admission rate, treatment compliance, OS, DFS and follow-up cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed lung cancer;
* Patients have received surgery, neoadjuvant therapy, adjuvant therapy, radiotherapy or other chemotherapy, such as cytotoxic chemotherapy, targeted therapy and immunotherapy;
* ECOG (Performance status) 0-1;
* Patients aged > 18 years and < 70 years;
* The patients themselves or their family members are familiar with mobile and internet;

Exclusion Criteria:

* Patients have disease progression in the screening period;
* Patients with symptomatic brain metastasis;
* Patients with dementia, schizophrenia or other psychological diseases that may affect the cognitive behavior;
* Other medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information;
* Women who are pregnant or in the period of breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
The quality of life after 6 months follow-up | From enrollment to 6 months after follow-up
  The evaluation of quality of life is based on FACT questionnaire (Version 4.0)

SECONDARY OUTCOMES:
The score of anxiety/depression after 6 months follow-up | From enrollment to 6 months after follow-up
  The evaluation of anxiety/depression is based on HADS questionnaire
The physical fitness score at the time of tumor progression | From enrollment to the time of tumor progression (up to 72 months)
  The physical fitness score at the time of tumor progression
The frequency of emergency treatment | 24 months after enrollment
  The frequency of emergency treatment
The frequency of rehospitalization | 24 months after enrollment
  The frequency of rehospitalization
The compliance of follow-up | 24 months after enrollment
  The evaluation of follow-up compliance is based on the frequency of drop out
Disease-free survival | 24 months after enrollment
Overall survival | 24 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The participant data will be encrypted and masked before uploading.

REFERENCES:
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Result] Dai W, Feng W, Zhang Y, Wang XS, Liu Y, Pompili C, Xu W, Xie S, Wang Y, Liao J, Wei X, Xiang R, Hu B, Tian B, Yang X, Wang X, Xiao P, Lai Q, Wang X, Cao B, Wang Q, Liu F, Liu X, Xie T, Yang X, Zhuang X, Wu Z, Che G, Li Q, Shi Q. Patient-Reported Outcome-Based Symptom Management Versus Usual Care After Lung Cancer Surgery: A Multicenter Randomized Controlled Trial. J Clin Oncol. 2022 Mar 20;40(9):988-996. doi: 10.1200/JCO.21.01344. Epub 2022 Jan 7. PMID 34995100